CLINICAL TRIAL: NCT03470714
Title: The Determination of Relationship Between Kinesiotaping and Contralateral Force Irradiation
Brief Title: Effect of Kinesiotaping on Force Irradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hdenizkulli
Record Dates: First submitted 2018-02-06; First posted 2018-03-20 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Force Irradiation; Kinesiotaping; EMG

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping Group (Experimental): The group in which kinesiotaping is applied to non-dominant biceps brachii muscle of participants before 24 hours the force irradiation experiment.
  Interventions: Other: Force Irradiation; Other: Kinesiotaping
- Control group (Active Comparator): The group in which the participants only perform the the force irradiation experiment.
  Interventions: Other: Force Irradiation

INTERVENTIONS:
Other: Force Irradiation — For the force irradiation, while the subjects perform dominant elbow flexion at an angular velocity of 60°/s for concentric contractions, 30°/s for eccentric contractions, at 90° elbow flexion position for isometric contractions with a maximal effort level, electrical activity of the non-dominant biceps brachii and triceps brachii muscles are recorded.
Other: Kinesiotaping — For kinesiotaping, the elbow positioned in 30°-45° flexion and kinesiotaping facilitation technique is applied origin to insertion of non-dominant biceps brachii muscle before 24 hours the experiment.
  Other Names: Force Irradiation
  Arms: Kinesiotaping Group

SUMMARY:
The study is assessed the electromyographic activity response of non-dominant biceps brachii muscle during unilateral-dominant concentric, eccentric and isometric biceps brachii muscle contractions under kinesiotaping and non-taping conditions. The aim of the study is to determine the synergistic effect of kinesiotaping which is applied on non-dominant biceps brachii muscle on force irradiation.

DETAILED DESCRIPTION:
Fourty healthy subjects with no history of neurological or recent musculoskeletal injury will participate the study.

Healthy subjects are arranged in two groups of stimulation: kinesiotaping group (kinesiotaping and force irradiation) and control group (only force irradiation). The electromyographic response of the resting arm (non-dominant) will be assessed during the dominant arm movement for all subjects. Additionally, in kinesiotaping group, kinesiotaping will be applied 24 hours before the experiment.

The electromyographic response of the resting arm will be assessed under three contraction type movement (isometric, eccentric and concentric contractions) The SEMG signals are analysed by using MATLAB®, suitable signal proccessing techniques (linear envelope, Root Mean Square etc) are chosed. The statistical analysis are done by using SPSS®, according to data distribution, "Independent Sample T Test" or "Mann-Whitney U Test" is utilized for comparing outcomes of control and KT groups.

ELIGIBILITY:
Inclusion Criteria:

* To be right-handed-dominant
* To have normal or corrected vision
* To have no formal history of any resistance training.

Exclusion Criteria:

* To have history of neurological or recent musculoskeletal injury

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Measurement of the surface electromyographic activity of left biceps brachii muscle by using surface electromyography device while the right elbow performs isometric elbow flexion | after inclusion
  while the right elbow performs isometric elbow flexion, electromyographic activity of left biceps brachii was determined by using surface electromyography device. After signal processing and normalization, the electromyographic data of kinesiotaping and control groups will be compared.
Measurement of the surface electromyographic activity of left triceps brachii muscle by using surface electromyography device while the right elbow performs isometric elbow flexion | after inclusion
  while the right elbow performs isometric elbow flexion, electromyographic activity of left triceps brachii was determined by using surface electromyography device. After signal processing and normalization, the electromyographic data of kinesiotaping and control groups will be compared.
Measurement of the surface electromyographic activity of left biceps brachii muscle by using surface electromyography device while the right elbow performs concentric elbow flexion. | after inclusion
  while the right elbow performs concentric elbow flexion, electromyographic activity of left biceps brachii was determined by using surface electromyography device. After signal processing and normalization, the electromyographic data of kinesiotaping and control groups will be compared.
Measurement of the surface electromyographic activity of left triceps brachii muscle by using surface electromyography device while the right elbow performs concentric elbow flexion | after inclusion
  while the right elbow performs isometric elbow flexion, electromyographic activity of left triceps brachii was determined by using surface electromyography device. After signal processing and normalization, the electromyographic data of kinesiotaping and control groups will be compared.
Measurement of the surface electromyographic activity of left biceps brachii muscle by using surface electromyography device while the right elbow performs eccentric elbow flexion | after inclusion
  while the right elbow performs eccentric elbow flexion, electromyographic activity of left biceps brachii was determined by using surface electromyography device. After signal processing and normalization, the electromyographic data of kinesiotaping and control groups will be compared.
Measurement of the surface electromyographic activity of left triceps brachii muscle by using surface electromyography device while the right elbow performs eccentric elbow flexion | after inclusion
  while the right elbow performs eccentric elbow flexion, electromyographic activity of left triceps brachii was determined by using surface electromyography device. After signal processing and normalization, the electromyographic data of kinesiotaping and control groups will be compared.

SECONDARY OUTCOMES:
Measurement of the electromyographic activity of left biceps brachii muscle during left elbow maximum isometric flexion by using electromyography device. | after inclusion
  Electromyographic activity of left elbow maximum isometric flexion is used for normalizing force irradiation data of left biceps brachii muscle
Measurement of the electromyographic activity of left triceps brachii muscle during left elbow maximum isometric extension by using electromyography device. | after inclusion
  Electromyographic activity of left elbow maximum isometric extension is used for normalizing force irradiation data of left triceps brachii muscle

CONTACTS AND LOCATIONS:
Overall Officials: Aydın AKAN, Study Director — Istanbul University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)